CLINICAL TRIAL: NCT05628974
Title: Normal Donor Blood Draws for Platelet Studies and Biomarker Evaluation (ND-PLT)
Acronym: ND-PLT
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Scott Cameron, MD, PhD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 20-413; 5R01HL158801-04 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center study at the Cleveland Clinic Main Campus designed to study biomarkers in healthy individuals to identify novel mechanisms of platelet activation and how platelets drive vascular inflammation and thrombosis in diseases.

DETAILED DESCRIPTION:
Our past studies have discovered novel platelet activation pathways that may be targets of therapeutic development. We have also defined an important role for a shift in platelet phenotype in vascular disease. Our studies use both in vivo animal models and validation using human platelets from isolated blood. Platelets from healthy individuals may be compared to patients with vascular diseases in the IRB approved protocol "Vascular Lab Resource" (IRB #19-1451) study which is actively recruiting patients at the Cleveland Clinic Main Campus and studies patients with vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years old
* Healthy Male & Female voluntary participants

Exclusion Criteria:

* Individuals who have taken anticoagulant or antiplatelet medications in past 10 days
* Individuals with hematopoetic diseases

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Voluntary donors will be screened by questioning for use of anti-coagulant medications such as aspirin or other non-steroidal anti-inflammatory agents, in the past 10 days, or for hematopoietic diseases. Only healthy volunteers included as platelet donors.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
To collect blood samples | 10 years
  To establish a biorepository for normal healthy cohort of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cameron, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laakso L. Migrants in hospital. Aust N Z J Obstet Gynaecol. 1973 Nov;13(4):231. doi: 10.1111/j.1479-828x.1973.tb02318.x. No abstract available. PMID 4532543
- [Background] [Hospital policy]. Rev Clin Inst Matern Lisb. 1965 Jul-Dec;16(62):59-70. No abstract available. Portuguese. PMID 5898983
- [Background] Lonnerdal B, Keen CL, Glazier CE, Anderson J. A longitudinal study of rhesus monkey (Macaca mulatta) milk composition: trace elements, minerals, protein, carbohydrate, and fat. Pediatr Res. 1984 Sep;18(9):911-4. doi: 10.1203/00006450-198409000-00023. PMID 6483513
- [Background] Faraday N, Goldschmidt-Clermont PJ, Bray PF. Gender differences in platelet GPIIb-IIIa activation. Thromb Haemost. 1997 Apr;77(4):748-54. PMID 9134654